CLINICAL TRIAL: NCT01325584
Title: Compassionate Use of Omegaven® in the Treatment of Parenteral Nutrition Induced Hepatic Injury
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Alternative product is now approved and available for use.
Sponsor: Midwestern Regional Medical Center (Other)
Responsible Party: Principal Investigator, Pankaj Vashi, MD, Lead National Medical Director, National Director Gastroenterology, Nutrition & Metabolic Support, Midwestern Regional Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRMC 10-06
Record Dates: First submitted 2011-03-25; First posted 2011-03-30 (Estimated); Results first posted 2018-06-27 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-07

CONDITIONS: Cancer; Hepatic Injury
MeSH Terms: conditions — Neoplasms | interventions — fish oil triglycerides; Fish Oils

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Omegaven (compassionate use) (Experimental): This is a compassionate use study. All participants will receive intravenous Omegaven (10% fish oil emulsion) with parenteral nutrition for 4 weeks.
  Interventions: Drug: Omegaven

INTERVENTIONS:
Drug: Omegaven — initial dose of 0.1 g/kg body weight (1ml/kg) and increased to 0.2 g/kg body weight (2ml/kg) on day 2 or 3 of treatment. The infusion rate will not exceed 0.5mL Omegaven/kg body weight/hr (corresponding to 0.05g fish oil/kg/hr). Patients will receive the initial infusion of PN containing Omegaven at Midwestern Regional Medical Center (MRMC) in the infusion center to observe for adverse reactions. Patients will continue to receive infusions at MRMC for the first 2 to 3 days of dosing. After tolerance is established, patients will receive treatment at home. All study patients will have a Screening Visit; Day 1, Day 2 and Day 3 visits; and weekly visits for one month.
  Other Names: fish oil

SUMMARY:
The purposes of this study are to make Omegaven® available to cancer patients with liver disease and to determine if Omegaven® can improve or prevent further liver disease. The study will also look at the effects Omegaven® has on immune function.

DETAILED DESCRIPTION:
This compassionate use study will include patients with advanced cancer requiring PN for long-term nutrition support who have developed PN-induced hepatic injury or who have existing hepatic dysfunction. Therapy with Omegaven will be provided at an initial dose of 0.1 g/kg body weight (1ml/kg) and increased to 0.2 g/kg body weight (2ml/kg) on day 2 or 3 of treatment. For patients > 120% ideal body weight, adjusted body weight will be used. The infusion rate will not exceed 0.5mL Omegaven/kg body weight/hr (corresponding to 0.05g fish oil/kg/hr). Omegaven will be co-administered via a y-site infusion, with containers being changed every 12 hours. The patient may receive other lipids to meet Essential Fatty Acid (EFA) and/or additional calorie needs. Patients will receive the initial infusion of PN containing Omegaven at Midwestern Regional Medical Center (MRMC) in the infusion center to observe for adverse reactions. If an adverse reaction is observed, IV steroids & benadryl will be administered & Omegaven will be discontinued. Patients will continue to receive infusions at CTCA for the first 2 to 3 days of dosing. After tolerance is established, patients will receive treatment at home with Coram. All study patients will have a Screening Visit; Day 1, Day 2 and Day 3 visits; and weekly visits for one month (see Table 2).

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female; ages 18 to 80 years old
2. Receiving treatment at Cancer Treatment Centers of America
3. Receiving PN (either in the infusion center or at home)
4. Have existing hepatic dysfunction defined as Elevation of > 3x the normal level of one or more of the following:Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), or Alanine Aminotransferase ALT) and/or Bilirubin > 2 mg/dl in the absence of biliary obstruction
5. Able to provide informed written consent

Exclusion Criteria:

1. Hypertriglyceridemia (triglycerides [TG] > 400)
2. Allergy to fish or egg protein
3. Currently on therapeutic doses of Coumadin, heparin, or low molecular eight heparin
4. Hemodynamically unstable
5. Bilirubin > 5 mg/dL
6. Documented liver metastases
7. Unstable diabetes with known diabetic ketoacidosis within 7 days of screening
8. Recent cardiac infarction (within 6 months) and taking plavix
9. Severe hemorrhagic disorders
10. Current anticoagulation therapy for deep venous thromboembolism or pulmonary embolism
11. Active sepsis
12. Undefined coma status
13. In patients with abnormal kidney function, renal insufficiency with calculated creatinine clearance < 30 mL/min
14. Pregnancy or lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-10; Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Vashi, MD, Principal Investigator — Midwestern Regional Medical Center
Locations (1):
- Cancer Treatment Centers of America at Midwestern Regional Medical Center, Zion, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
At present, no plan to share individual participant data.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omegaven (Compassionate Use)
Started | 12
Completed | 11
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Omegaven (Compassionate Use)
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Maximum Conjugated Bilirubin
Description: Highest detected lab values will be summarized between baseline and end of study participation.
Time Frame: Assessed at day 1, 2, 3, and weekly therafter, up to 4 weeks.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Omegaven (Compassionate Use)
Number analyzed (Participants) | 11
mg/dl | 1.0 (0.1)

2. Primary Outcome: Average Change in Alkaline Phosphatase
Description: lab values will be summarized at baseline and as change from baseline to worst follow-up value.
Time Frame: Assessed at day 1, 2, 3, and weekly therafter, up to 4 weeks.
Population: Average Improvement in Alkaline Phosphatase
Measure: Mean (Full Range); unit: U/L
Arm/Group | Omegaven (Compassionate Use)
Number analyzed (Participants) | 11
U/L
  Baseline | 457.6 [390 to 1006]
  4 Week Nadir | 360.4 [193 to 723]
Statistical Analysis 1: Comparison: Omegaven (Compassionate Use); Test type: Superiority; p = .07, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Number of Patients Experiencing Adverse Events
Description: The number of patients reporting or experiencing adverse effects will be reported.
Time Frame: Assessed at day 1, 2, 3, and weekly therafter, up to 4 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Omegaven (Compassionate Use)
Number analyzed (Participants) | 11
Participants | 1

4. Primary Outcome: Average Improvement in AST
Description: Lab values will be summarized at b aselin4e and as change from baseline to worst follow-up value.
Time Frame: Assessed at day 1, 2, 3, and weekly therafter, up to 4 weeks.
Measure: Mean (Full Range); unit: U/L
Arm/Group | Omegaven (Compassionate Use)
Number analyzed (Participants) | 11
U/L
  Baseline | 88.7 [31 to 402]
  4 Weeks Nadir | 69.9 [24 to 160]
Statistical Analysis 1: Comparison: Omegaven (Compassionate Use); Test type: Superiority; p = .53, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Average Improvement in ALT
Description: Laboratory values will be summarized at baseline and as change from baseline to worst follow-up value
Time Frame: Assessed at day 1, 2, 3, and weekly therafter, up to 4 weeks.
Measure: Mean (Full Range); unit: U/L
Arm/Group | Omegaven (Compassionate Use)
Number analyzed (Participants) | 11
U/L
  Baseline | 133.6 [29 to 456]
  4 Weeks Nadir | 101.4 [15 to 336]
Statistical Analysis 1: Comparison: Omegaven (Compassionate Use); Test type: Superiority; p = .48, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Omegaven (Compassionate Use)
All-Cause Mortality (participants affected / at risk) | 1/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omegaven (Compassionate Use) (N=11)
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2011-02-04): https://cdn.clinicaltrials.gov/large-docs/84/NCT01325584/Prot_000.pdf